CLINICAL TRIAL: NCT04874909
Title: Classification and Functional Stratification of the Patients With Ciliopathy and Identification of Biomarkers to Improve Their Prognosis
Brief Title: Classification, Functional Stratification and Biomarkers in Ciliopathy (CILLICORIRCM)
Acronym: CILLICORIRCM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP200896; ID-RCB Number (Other: 2020-A02356-33)
Record Dates: First submitted 2021-03-31; First posted 2021-05-06 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Ciliopathies; Nephronophthisis; Senior-Loken Syndrome; Joubert Syndrome; Jeune Syndrome; Bardet-Biedl Syndrome
Keywords: Ciliopathies; Pediatrics; Genetic diseases; Chronic Kidney Disease; Biomarkers
MeSH Terms: conditions — Ciliopathies; Nephronophthisis, familial juvenile; Senior Loken Syndrome; Agenesis of Cerebellar Vermis; Jeune syndrome; Bardet-Biedl Syndrome; Genetic Diseases, Inborn; Renal Insufficiency, Chronic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- "Case" Patient (Other): Patient with ciliopathy
  Interventions: Other: Blood sample; Other: Urine sample
- Healthy related individual (Other): Individual without ciliopathy but related to a patient with ciliopathy (father, mother, brother, sister)
  Interventions: Other: Blood sample; Other: Urine sample
- "Negative Control" patient (Other): patient without renal disease
  Interventions: Other: Blood sample; Other: Urine sample
- "Positive Control" patient (Other): patient with renal disease other that ciliopathy but with a similar renal function to the ciliopathy group ("case" patient)
  Interventions: Other: Blood sample; Other: Urine sample

INTERVENTIONS:
Other: Blood sample — Blood sample of 15ml max by subject (case, related individual, control) once time:
  * subject less than 5 kg : 1.8 to 4.5 ml max
  * subject 5 kg to 10 kg : 4.5 to 9 ml max
  * subject 10 kg to 15 kg : 9 to 13.5 ml
  * subject 15 kg to 20 kg : 13.5 to 15 ml max
Other: Urine sample — Urine sample (500 ml) once time

SUMMARY:
The purpose of the C'IL-LICO RICM study is to develop innovative and transformative diagnostic and prognostic for patients suffering from ciliopathies leading to renal failure.

The objectives is to decipher disease mechanisms and highlight signaling pathways altered in at-risk to develop renal failure patient groups and to produce a prognostic biomarker-based kit to predict the evolution of ciliopathy patients towards renal impairment.

DETAILED DESCRIPTION:
Ciliopathies are a large group of rare and severe genetic diseases caused by ciliary dysfunction, in which nearly all organs can be affected. In spite of being individually rare, they affect collectively up to one per 2000 people. Over the past two decades, more than 90 genes have been reported as mutated in ciliopathy patients. Most proteins encoded by these genes play key roles in the biogenesis or function of cilia, in which they define different functional subdomains. Genetic analyses of ciliopathies revealed a vast clinical variability and a broad genetic heterogeneity as: 1) mutations of the same disease-causing gene can result in distinct clinical entities and, conversely, 2) mutations in several independent genes can lead to similar clinical features, implying both phenotypic and genetic overlaps. The extent and severity of organ involvement may be correlated in part with the nature or location of the mutational event, the cell/tissue specific expression and effect of the mutated protein on cilia dysfunction.

Renal involvement is one of the most frequent manifestations in ciliopathies, and it leads to excessive morbidity and mortality. This includes renal cystic dysplasia (RCD), a kidney developmental defect, and nephronophthisis (NPHP), a chronic tubulointerstitial nephritis, both disorders representing frequent causes of end-stage renal disease (ESRD) during childhood to early adulthood. This makes ESRD a terminal endpoint of either isolated or syndromic ciliopathies, with, hitherto, no available curative treatment of chronic kidney disease whatsoever. The only bearable option is renal transplantation. As the average life-span of a functioning kidney transplant is about 10-15 years, it is urgent to identify therapeutic solutions that slow down progression of CKD in ciliopathies, and delay or avoid dialysis or transplantation. Today, the diagnosis of ciliopathies is first based on primary clinical manifestations, and then confirmed by gene mutation identification. However, even in patients with identified causative mutations, it is impossible to predict the severity of the disease, the risk of appearance (if not present at diagnosis), and/or the rate of progression of CKD. Thus, a crucial issue in the field of ciliopathies is to be able to perform early detection of at-risk patients prior to development of CKD as well as to predict disease progression rate.

ELIGIBILITY:
Inclusion Criteria:

"Case" Patient :

* with nephronophthisis or ciliopathy with known genetic diagnosis or not
* signed the Informed consent form (patient or legal guardians if minor/incapable major)
* no limit of age, this patients could be recruited from the birth
* social insurance affiliation

Healthy related individual :

* related with a included patient (father, mother, brother, sister)
* signed the Informed consent form (major or legal guardians if minor/incapable major)
* no limit of age, this patients could be recruited from the birth
* social insurance affiliation

"Negative Control" patient :

* without chronic renal failure
* signed the Informed consent form (major or legal guardians if minor/incapable major)
* no limit of age, this patients could be recruited from the birth
* social insurance affiliation

"Positive Control" patient :

* with chronic renal failure not related with a ciliary dysfunction
* signed the Informed consent form (major or legal guardians if minor/incapable major)
* no limit of age, this patients could be recruited from the birth
* social insurance affiliation

Exclusion Criteria "Case" Patient :

* pregnant, parturious and nursing mothers.
* with functional renal graft
* use an experimental treatment during 30 days before inclusion date

Healthy related individual :

- pregnant, parturious and nursing mothers.

"Negative Control" patient :

- pregnant, parturious and nursing mothers.

"Positive Control" patient :

* pregnant, parturious and nursing mothers.
* with functional renal graft
* use an experimental treatment during 30 days before inclusion date

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-11-08 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Change in transcriptional profiles in different subtypes of ciliopathy patients and control subjects | 3 years
  RNA-sequencing analysis will be utilized to identify changes in transcriptional profiles and biological pathways in subgroups of patients to research whether the target mutation gene combination analyzed by transcription group was consistent with clinical cell morphological diagnosis and disease progression.
  Different human models will be used: Urine-derived Renal Epithelial Cells (URECs), renal organoids from patients derived induced Pluripotent Stem Cells (iPSCs) and urines.

SECONDARY OUTCOMES:
Change in proteome profiles in different subtypes of ciliopathy patients and control subjects | 3 years
  Proteomics analysis will be utilized to identify changes in proteome profiles in subgroups of patients to research whether the target mutation gene combination analyzed by proteomics group was consistent with clinical cell morphological diagnosis and disease progression.
  Different human models will be used: Urine-derived Renal Epithelial Cells (URECs), renal organoids from patients derived induced Pluripotent Stem Cells (iPSCs) and urines.
Change in metabolome profiles in different subtypes of ciliopathy patients and control subjects | 3 years
  Metabolomics analysis will be utilized to identify changes in metabolome profiles in subgroups of patients to research whether the target mutation gene combination analyzed by metabolomics group was consistent with clinical cell morphological diagnosis and disease progression.
  Different human models will be used: Urine-derived Renal Epithelial Cells (URECs), renal organoids from patients derived induced Pluripotent Stem Cells (iPSCs) and urines.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie SAUNIER, PhD, Study Chair — Imagine Institute
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No